CLINICAL TRIAL: NCT00780286
Title: Retention of an Orally Administered Investigational Device vs Commerical Device in the Oral Cavity and Oropharynx of Healthy Human Male Volunteers
Brief Title: Evaluate Retention of an Orally Administered Device Using Gamma Scintigraphy Study 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008068
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Polymer based lubricating liquid
- 2 (Active Comparator)
  Interventions: Device: Moi-Stir

INTERVENTIONS:
Device: Polymer based lubricating liquid — 5 mls of radiolabeled polymer blend of carboxymethylcellulose, polyoxyl 40 stearate, and polyethylene oxide that coats and protects the mucus membrane
  Arms: 1
Device: Moi-Stir — 2 sprays (0.35 mL) of the radiolabeled commercial device. A blend of Water, sorbitol, carboxymethylcellulose, sodium, methylparaben, propylparaben, potassium chloride, dibasic sodium phosphate, calcium chloride, magnesium chloride, sodium chloride, flavor.
  Arms: 2

SUMMARY:
Single usage, open label study in up to 40 adult healthy males. Eligible subjects will receive a single usage of the investigational or commercial device. Retention of the radiolabeled device will be monitored using gamma scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Refrain from nasal, throat, or lung inhalants and exercise for 24 hour prior to the test
* Are able to tolerate the procedure and
* Be generally healthy

Exclusion Criteria:

* Have history of allergy or hypersensitivity to the study ingredients
* Major diseases
* Taking medication regularly
* Radiation exposure recently

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Area under the curve for volume of investigational device retained in the oral cavity. | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Walter J Doll, PhD, RPh, Principal Investigator — Scintipharma, Inc
Locations (1):
- Walter J Doll, PhD, RPh, Lexington, Kentucky, United States